CLINICAL TRIAL: NCT06663150
Title: Effectiveness of a Health Intervention With a Socio-community Approach on Frailty in Older Adults With Pre-frailty
Brief Title: Effectiveness of a Socio-Community Health Intervention on Pre-Frailty in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keralty SAS. Colombia (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 092-24 UNV
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Frail Elderly Syndrome
Keywords: Prefrailty; Frailty; Older Adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Education Component: Lectures and workshops aimed at enhancing awareness and personal growth through knowledge and emotional reflection.
  Cognitive Component: One-hour sessions divided into introduction (15 min), cognitive stimulation activities (35 min), and closure with reflection and a brief survey.
  Physical Activity Component: A 10-minute warm-up, followed by 30 minutes of guided exercises for balance, coordination, and strength, ending with a 10-minute cool-down.
  Nutrition Component: Practical workshops focused on healthy eating, including menu planning and food preparation.
  Socio-Community and Occupational Component: Encourages community integration and social networking, with gardening activities for growing herbs and vegetables.
  Autonomous Activities: Participants implement physical activity recommendations in daily life, with weekly follow-ups by the research team using the RedCap platform for monitoring.
  Interventions: Behavioral: health intervention with a socio-community approach
- Control group (No Intervention): The control group will maintain the usual care provided by their healthcare service provider.

INTERVENTIONS:
Behavioral: health intervention with a socio-community approach — The intervention consists of five components, including education, cognitive stimulation, physical activity, nutrition, and socio-community aspects. The duration of the intervention will be 6 months and will be conducted in either in-person or virtual format, individually or in groups, depending on the nature of each component. Mode of Delivery:
  The intervention will be offered in both in-person and synchronous virtual formats. Participants who are unable to attend in person or who face difficulties doing so on any occasion will have the option to join the sessions through a real-time videoconferencing platform. In both modalities, the professionals in charge will supervise and guide the activities, ensuring proper execution and adherence to the study's objectives. The research team will maintain a detailed record of attendance and participation using the RedCap platform for appropriate tracking.
  Arms: Experimental group

SUMMARY:
The objective of this study is: To evaluate the effectiveness of a health intervention with a socio-community approach on frailty in older adults with pre-frailty.

Specific Objectives:

To characterize the study population according to sociodemographic and clinical variables.

To evaluate the effect of the intervention on the functionality domain at 3 and 6 months.

To evaluate the effect of the intervention on the cognitive-emotional domain at 3 and 6 months.

To evaluate the effect of the intervention on the socio-community domain at 3 and 6 months.

To evaluate the effect of the intervention on frailty in older adults. To determine the proportion of participants hospitalized during the study period.

To determine the proportion of participants who visited the emergency room during the study period.

To determine the proportion of participants in long-term care facilities. To determine the proportion of adverse events associated with the intervention.

Study Hypothesis

The mean frailty score pre-intervention is equal to the mean frailty score post-intervention.

The mean frailty score pre-intervention is different from the mean frailty score post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 60 years old classified as pre-frail in the last 3 months and documented in their medical history.
* Individuals who meet the requirements and provide voluntary informed consent for their participation.
* Individuals available to remain in Bogotá D.C. during the study period.

Exclusion Criteria:

* Individuals receiving care at community-focused medical centers.
* Individuals attending community dining programs, physical activity programs, community groups, care blocks, volunteering, or other related activities.
* Individuals who have experienced falls in the last 6 months with clinical consequences (hospitalization, fractures, traumatic brain injury).
* Individuals with a clinical history of moderate cognitive impairment, neurodegenerative diseases (e.g., Parkinson's disease), and/or neuro-musculoskeletal disorders, active cancer, end-stage renal disease, unstable ischemic heart disease, uncontrolled arrhythmias, severe aortic stenosis, uncontrolled hypertension (>180/100 mmHg), or advanced heart failure, exacerbation of chronic diseases (COPD, heart failure), unrehabilitated severe hearing loss, deafness, or blindness with communication limitations.
* Acute conditions requiring hospitalization, such as acute myocardial infarction or urinary tract infections.
* Bone fractures in the last 3 months.
* Individuals unable to follow instructions or with behavioral changes that hinder their participation in the study.
* Individuals with severe psychiatric illness that, in the physician's judgment, prevents proper adherence to the study intervention.
* Institutionalized individuals in long-term care facilities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Score on the FRAIL Scale | Baseline, 3, 6 Months
  Frailty will be assessed using the FRAIL Scale, which evaluates five domains: fatigue, resistance, ambulation, illnesses, and weight loss. The total score ranges from 0 to 9, where higher scores indicate greater frailty

SECONDARY OUTCOMES:
Barthel Index | Baseline, 3, 6 Months
  Measures independence in basic activities of daily living. The score ranges from 0 to 100, where higher scores indicate greater independence.
Lawton Score | Baseline, 3, 6 Months
  Assesses instrumental activities of daily living (IADLs), with a score range of 0 to 8. Higher scores indicate better ability to perform IADLs independently.
Downton Scale | Baseline, 3, 6 Months
  Evaluates the risk of falls in older adults, considering factors such as previous falls, medication use, sensory deficits, mental status, and walking ability. The score ranges from 0 to 14, where higher scores indicate a higher risk of falls.
Score on the Montreal Cognitive Assessment (MoCA) | Baseline, 3, 6 Months
  The MoCA is a global cognitive screening tool that assesses memory, attention, language, abstraction, executive function, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function
Score on the Yesavage Geriatric Depression Scale (GDS) | Baseline, 3, 6 Months
  The GDS is a tool used to assess depression in older adults, with scores ranging from 0 to 15. Higher scores indicate more severe depression.
Score on the Gijón Family-Social Assessment Scale | Baseline, 3, 6 Months
  The Gijón Family-Social Assessment Scale evaluates the socio-family situation of the patient, considering factors such as economic situation, family relationships, and social support. The score ranges from 0 to 15, with higher scores indicating greater socio-family vulnerability
Score on the Lubben Social Network Scale | Baseline, 3, 6 Months
  The Lubben Social Network Scale assesses the social support and contact network of an individual, with a score range of 0 to 30. Higher scores indicate a stronger social support network.
Health-Related Quality of Life Measured by EQ-5D-3L | Baseline, 3, 6 Months
  The EQ-5D-3L is a health-related quality of life measurement tool that consists of two parts: a descriptive system covering five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a Visual Analogue Scale (VAS) where participants rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health). The descriptive system generates a health profile, and the VAS provides a quantitative measure of perceived overall health.
Number of Hospital Admissions | During the 6-month intervention
  The total number of hospital admissions recorded during the 6-month intervention period.
Total Number of Hospitalization Days | During the 6-month intervention
  The total number of days spent in the hospital, summing all admissions during the 6-month intervention period.
Total Number of Emergency Room Admissions | During the 6-month intervention.
  The total number of emergency room admissions recorded during the 6-month intervention period.
Requirement for Admission to Long-Term Care Facilities | During the 6-month intervention.
  This measure tracks whether participants require admission to long-term care facilities during the 6-month intervention period.
Utilization of Social Health Assets | During the 6-month intervention.
  This measure tracks the use of social health services, including community-based resources,

OTHER OUTCOMES:
Adverse Events | During the 6-month intervention.
  Adverse events refer to any undesirable experiences or occurrences resulting from the intervention, including but not limited to side effects, complications, or unexpected outcomes. All adverse events will be recorded and categorized based on their severity (e.g., mild, moderate, severe) and their relationship to the intervention (e.g., related, possibly related, unrelated)

CONTACTS AND LOCATIONS:
Overall Officials: Lina Sofía Morón-Duarte, PhD, Study Chair — keralty

IPD SHARING:
Plan to Share IPD: No